CLINICAL TRIAL: NCT04630444
Title: An Investigational Study of Riluzole Effects on Hippocampus Biomarkers
Brief Title: Riluzole Effects on Hippocampus Biomarkers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Isabelle Rosso, Associate Professor, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P002687
Record Dates: First submitted 2017-07-14; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Group (Experimental): 30 PTSD patients receiving riluzole 100 mg daily (50 mg bid).
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole — 30 PTSD patients with riluzole 100 mg daily (50 mg bid).

SUMMARY:
To examine the clinical efficacy of the anti-glutamatergic medication riluzole in posttraumatic stress disorder (PTSD), and its effect on hippocampus biomarkers that our laboratory previously has identified using MRS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18-65.
2. Right handed
3. Able to provide written informed consent.
4. Meets DSM-5 criteria for PTSD (current month and past 3 months).
5. If already receiving psychiatric intervention(s), must be on a stable regimen.
6. Has normal physical examination, laboratory test results, and electrocardiogram results at pre-treatment visit.

Exclusion Criteria:

1. Unwillingness or inability to provide written informed consent.
2. Unable to swallow pills.
3. Unable to tolerate blood draws.
4. Currently enrolled in another intervention study.
5. Imminent risk for self-harm (assessed by a licensed clinician)
6. Active psychotic symptoms.
7. Current panic disorder.
8. Lifetime history of schizophrenia spectrum disorder, bipolar disorder, obsessive compulsive disorder, anorexia nervosa, seizure disorder, or neurologic disorder.
9. Urine toxicology positive for drug(s) of abuse.
10. Evidence of any clinically significant medical disease.
11. Women who test positive for ß-HCG, self-report as pregnant, or are nursing.
12. Substance or alcohol abuse within 3 months of Visit 1. Substance or alcohol dependence within 6 months of Visit 1.
13. Excessive caffeine use, defined as regular consumption of >700mg caffeine per day.
14. Treatment with an antipsychotic, valproate, other anticonvulsant, reversible MAOI within 4 weeks of Visit 1. Other excluded medications will be those with (1) known glutamatergic effects, (2) previous MRS evidence of effects on brain glutamate, (3) potential effects on riluzole levels or (4) risk of neutropenia - used within 4 weeks of the first study visit.
15. Previous exposure to riluzole or ketamine.
16. Treatment with any investigational medicine within 30 days of Visit 1.
17. Treatment with electroconvulsive therapy (ECT) within 3 months of Visit 1.
18. Uncorrected thyroid disease.
19. Any screening laboratory assay that is deemed to be a clinically significant abnormality by the investigator, with the exception of liver function tests (AST, ALT, alkaline phosphatase), which must be within 1.5 times the upper limit of normal.
20. Any contraindications to having an MRI scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
Assessing the clinical efficacy of riluzole in PTSD | weeks 1-8
  Testing the hypothesis that riluzole monotherapy will yield within-subject reductions in PTSD total symptoms (CAPS total score)
Assessing the clinical efficacy of riluzole in PTSD | weeks 1-8
  Testing the hypothesis that riluzole monotherapy will yield within-subject reductions in PTSD intrusion symptoms (CAPS intrusion subscale)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided